CLINICAL TRIAL: NCT02958176
Title: Autonomic Imbalance and Female Sexual Arousal Disorder: The Identification of Heart Rate Variability Level as a Risk Factor and Treatment Target
Brief Title: Heart Rate Variability Biofeedback for Female Sexual Arousal Disorder
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Texas at Austin (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2016-08-0074
Record Dates: First submitted 2016-10-31; First posted 2016-11-08 (Estimated); Last update posted 2018-10-11 (Actual); Status verified 2018-10

CONDITIONS: Female Sexual Arousal Disorder
MeSH Terms: interventions — Autogenic Training

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (3):
- HRV Biofeedback (Experimental): At home HRV biofeedback using mobile device
  Interventions: Behavioral: HRV Biofeedback
- HRV Biofeedback with Autogenic Training (Experimental): At home HRV biofeedback using mobile device plus autogenic training recording
  Interventions: Behavioral: HRV Biofeedback; Behavioral: Autogenic Training
- Wait List (No Intervention): Wait list control

INTERVENTIONS:
Behavioral: HRV Biofeedback — At-home heart rate variability biofeedback using Elite HRV app and Polar H7 chest strap
  Arms: HRV Biofeedback; HRV Biofeedback with Autogenic Training
Behavioral: Autogenic Training — Autogenic training recording provided on a CD
  Arms: HRV Biofeedback with Autogenic Training

SUMMARY:
Low resting heart rate variability (HRV) has been associated with sexual arousal problems and overall sexual dysfunction in women. Research has indicated that HRV biofeedback leads to increases in HRV as well as improvements in symptoms associated with several psychological disorders, some of which are comorbid with sexual arousal problems in women. Autogenic training also facilitates increases in HRV and was recently associated with acute increases in sexual arousal among sexually healthy women. The primary aim of the current study is to examine the efficacy of HRV biofeedback, with and without autogenic training, for the treatment of female sexual arousal disorder (FSAD).

DETAILED DESCRIPTION:
Women who meet ICD-10-CM diagnostic criteria for FSAD will be recruited and randomized into one of three conditions, HRV biofeedback (n = 25), HRV biofeedback plus autogenic training (n = 25), or wait-list control (n = 15). All participants will complete a baseline assessment, during which their resting state HRV and vaginal pulse amplitude (VPA) will be measured. The participants in the two biofeedback conditions will receive training in HRV biofeedback from the experimenter, and they will be provided with the materials necessary to guide self-practice in HRV biofeedback at home. Participants in these two conditions will be instructed to engage in at-home HRV biofeedback (with or without autogenic training) at least 5 times over a period of two weeks, during which they will report levels of arousal in a sexual activity diary. Participants in the wait-list control condition will report levels of arousal in a sexual activity diary. After two weeks, participants in all three conditions will return to the laboratory, where their physiological and psychological sexual arousal will be measured. Over the next two weeks, participants in the two biofeedback conditions will be asked to complete 5 more self-guided biofeedback sessions along with the sexual activity diary. Participants in all three conditions will return to the lab for a final assessment to measure post-treatment HRV and VPA levels as well as psychological sexual arousal. To our knowledge, this study will be the first randomized controlled trial of HRV biofeedback in women with sexual arousal problems. If the intervention increases arousal in this population, this study may offer a promising cost-effective psychosocial treatment for women with sexual arousal problems.

ELIGIBILITY:
Inclusion Criteria:

* Premenopausal (18-40 years)
* Fluent in English
* Heterosexual or bisexual
* Score of 26.55 or less on the Female Sexual Function Index (FSFI)
* Current sexual arousal dysfunction
* Ownership of an Elite HRV compatible device (recent iPhone, iPad, or Android)

Exclusion Criteria:

* Pregnant or breastfeeding
* History of or current sexually transmitted infections
* History of major pelvic surgery
* History of childhood sexual abuse
* Currently taking androgens, estrogens, or other medical treatments to enhance sexual arousal
* Current psychosis
* If on antidepressants or antihypertensives, must be stabilized for at least 3 months

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 65 (Actual)
Dates: Start 2016-10; Primary Completion 2018-01 (Actual); Study Completion 2018-01 (Actual)

PRIMARY OUTCOMES:
Physiological sexual arousal assessed by vaginal photoplethysmography | One month
Subjective sexual arousal assessed by Film Scale (Heiman & Rowland, 1983) | One month
Sexual function assessed by Female Sexual Function Index (Rosen et al., 2000) | Two months

SECONDARY OUTCOMES:
Depression symptoms assessed by Beck Depression Inventory-II (Beck, Brown, & Steer, 1996) | Two months
Anxiety symptoms assessed by Beck Anxiety Inventory (Beck et al., 1988) | Two months
Interoceptive awareness assessed by the Multidimensional Assessment of Interoceptive Awareness (Mehling et al., 2012) | Two months

CONTACTS AND LOCATIONS:
Overall Officials: Cindy M Meston, Principal Investigator — The University of Texas at Austin
Locations (1):
- The University of Texas at Austin, Austin, Texas, United States

IPD SHARING:
Plan to Share IPD: Undecided